CLINICAL TRIAL: NCT01904630
Title: Exom-sekvensering for å Identifisere høyrisiko Genvarianter i en Familie Predisponert for Colorectal Cancer
Brief Title: Sequencing to Identify Gene Variants in Familial Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/1707
Record Dates: First submitted 2013-04-23; First posted 2013-07-22 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer
Keywords: gene sequencing; familial; risk factors
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples for DNA sequencing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CRC high risk: Participants belong to a family with increased risk for CRC, will be analyzed with gene sequencing
  Interventions: Genetic: gene sequencing

INTERVENTIONS:
Genetic: gene sequencing — Gene sequencing by exome capture and high throughput sequencing for identification of rare variants

SUMMARY:
The project will use exome sequencing to search for genetic predispositions for familial colorectal cancer (CRC). Except for certain syndromes there is today no good method for identifying individuals with a hereditary high risk for CRC (about 25% of the cases). There is currently no routine screening of the population in Norway for CRC today. Coloscopy, which is the most reliable method, is demanding with respect to resources, it can be painful, and may have complications. This project will attempt to find genetic determinants for identification of individuals with increased risk for familial CRC. Such methods will reduce unnecessary medical examination of unaffected family members, and will make it easier to focus health services on individuals with increased risk. This will represent a significant contribution towards improved health reduced death rate caused by CRC. The project includes research on the ethical aspects, in particular challenges related to how feedback to donors is handled.

DETAILED DESCRIPTION:
Participants will be from a specific family, and will be selected by invitation to volunteer.

ELIGIBILITY:
Inclusion Criteria:

* Member of a specific family with increased risk of CRC, including individuals both with and without CRC

Exclusion Criteria:

* Young age

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A specific family showing increased risk for CRC
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2012-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Data on association between sequence variants in exons and CRC risk | Data available within 18 months after recruitment completed
  For each participant the genome will be analyzed by exome capture and high throughput sequencing. The exome data will be compared between participants and to reference data for identification of unique variants that can be associated with disease risk.

CONTACTS AND LOCATIONS:
Overall Officials: Finn Drabløs, PhD/Prof, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Hansen MF, Johansen J, Bjornevoll I, Sylvander AE, Steinsbekk KS, Saetrom P, Sandvik AK, Drablos F, Sjursen W. A novel POLE mutation associated with cancers of colon, pancreas, ovaries and small intestine. Fam Cancer. 2015 Sep;14(3):437-48. doi: 10.1007/s10689-015-9803-2. PMID 25860647